CLINICAL TRIAL: NCT00821691
Title: Action of the Amantadine on Post Stroke Aphasic Patients' Language and Communication
Brief Title: Action of Amantadine on Post-Stroke Aphasic Patients
Acronym: CELIC-1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 01-APN-08
Record Dates: First submitted 2009-01-09; First posted 2009-01-13 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2013-06

CONDITIONS: Cerebral Infarction
Keywords: cerebral infarction
MeSH Terms: conditions — Cerebral Infarction | interventions — Amantadine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Amantadin - Placebo: 5 amantadin caps - 4 days wash out - 5 placebo caps
  5 amantadin caps (100mg); 2 caps a day during 3 days; after wash out period (4 days): 5 placebo caps (2 caps a day during 3 days)
  Interventions: Drug: Amantadin; Drug: Placebo
- 2 (Other): Placebo - Amantadin: 5 placebo caps - 4 days wash out - 5 amantadin caps
  5 placebo caps: 2 caps a day during 3 days after wash out period (4 days): 5 amantadin caps(100mg) (2 caps a day during 3 days)
  Interventions: Drug: Amantadin; Drug: Placebo

INTERVENTIONS:
Drug: Amantadin — Amantadin caps
Drug: Placebo — Placebo caps

SUMMARY:
The objective of the study is to test the action of the amantadine, as DOPA-agonist, in a double blind cross-over trial, amantadine / placebo, on the verbal fluency of chronic post stroke aphasic patients.

DETAILED DESCRIPTION:
In France, there are around 30000 aphasic patients. The actual taking care of these patients after stroke includes the treatment of acute stage in stroke unit, followed by rehabilitation program. However, most non fluent aphasic patients remain chronically handicapped despite of intensive logopedic training.

The objective of this clinical project is to test the action of pharmacologic agents on verbal fluency of aphasic patients victims of cerebral infarctions. Only a few studies have been done with various pharmacologic agents, and although the results were not clearly conclusive, they were sufficiently positive for suggesting to launch a well controlled randomized cross-over study.

Then the objective of study is to test the action of the amantadine, as DOPA-agonist, in a double blind cross-over trial, amantadine / placebo, on the verbal fluency of chronic post stroke aphasic patients.

ELIGIBILITY:
Inclusion Criteria:

* RANKIN < 3
* > 18 years and < 75
* francophone
* within cognitive deficit known before stroke
* stroke, single in sylvian artery area
* aphasia " non fluent " following a stroke
* stroke > six month
* stable treatment

Exclusion Criteria:

* RANKIN > 3
* non francophone
* do not read nor write
* many stroke - against indication
* participated in another clinical trial
* deaf or blind
* intercurrent disease
* new treatment (< 2 months) cognitive
* pregnant or lactating

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Confirm that the possibility of significantly improving the verbal fluency and communication of patients with "not fluent" aphasia at the chronic stage when logopedic rehabilitation is "stabilized" (> 6months). | 2 years

SECONDARY OUTCOMES:
Codify a drug test to be included in the" recommendations "to take care of these patients | 2 years
Establish correlations between clinical, neuroradiological lesions and pharmacological responses, as to argue in favour of long-term treatment | 2 years
Identify extra linguistic components of communication influenced by amantadine | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Marcel CHATEL, MDPH, Principal Investigator — University hospital of Nice; Hélène MAHAGNE, PH, Study Director — University hospital of Nice; Sylvain LACHAUD, PH, Study Director — University hospital of Nice
Locations (6):
- France (6):
  - CH Saint Pierre La Réunion, Saint-Pierre, Ile de La Réunion
  - University hospital of Bordeaux, Bordeaux
  - CHU de Dijon, Dijon
  - CHU Limoges, Limoges
  - CHU de Nice, Nice
  - CHU Rennes, Rennes